CLINICAL TRIAL: NCT03089112
Title: A Randomized, Open-label, Crossover Study to Investigate the Pharmacokinetic Drug Interactions and the Safety Between HGP1607 and HGP1501 in Healthy Male Volunteers
Brief Title: Pharmacokinetic Drug Interactions Between HGP1607 and HGP1501
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-BAVI-101
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Seguence 1 (Experimental): Period 1 : HGP1607 Period 2 : HGP1501 Period 3 : HGP1607+HGP1501
  Interventions: Drug: HGP1607; Drug: HGP1501; Drug: HGP1607+HGP1501
- Seguence 2 (Experimental): Period 1 : HGP1607 Period 2 : HGP1607+HGP1501 Period 3 : HGP1501
  Interventions: Drug: HGP1607; Drug: HGP1501; Drug: HGP1607+HGP1501
- Seguence 3 (Experimental): Period 1 : HGP1501 Period 2 : HGP1607 Period 3 : HGP1607+HGP1501
  Interventions: Drug: HGP1607; Drug: HGP1501; Drug: HGP1607+HGP1501
- Seguence 4 (Experimental): Period 1 : HGP1501 Period 2 : HGP1607+HGP1501 Period 3 : HGP1607
  Interventions: Drug: HGP1607; Drug: HGP1501; Drug: HGP1607+HGP1501
- Seguence 5 (Experimental): Period 1 : HGP1607+HGP1501 Period 2 : HGP1607 Period 3 : HGP1501
  Interventions: Drug: HGP1607; Drug: HGP1501; Drug: HGP1607+HGP1501
- Seguence 6 (Experimental): Period 1 : HGP1607+HGP1501 Period 2 : HGP1501 Period 3 : HGP1607
  Interventions: Drug: HGP1607; Drug: HGP1501; Drug: HGP1607+HGP1501

INTERVENTIONS:
Drug: HGP1607 — Take it once per period
Drug: HGP1501 — Take it once per period
Drug: HGP1607+HGP1501 — Take it once per period

SUMMARY:
A Randomized, Open-label, Crossover Study to Investigate the Pharmacokinetic drug interactions and the Safety between HGP1607 and HGP1501 in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* 1.age 19~40 years
* 2.The result of BMI is not less than 19 kg/m2 , no more than 28 kg/m2
* 3.Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
AUClast of HGP1607 | 16, -12, -8, 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96,120h
Cmax of HGP1607 | 16, -12, -8, 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96,120h
baseline corrected AUClast of HGP1501 | 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72, 96,120h
baseline corrected Cmax of HGP1501 | 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72, 96,120h

SECONDARY OUTCOMES:
AUCinf of HGP1607 | 16, -12, -8, 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96,120h
Tmax of HGP1607 | 16, -12, -8, 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96,120h
T1/2 of HGP1607 | 16, -12, -8, 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 24, 48, 72, 96,120h
AUClast of HGP1501 | 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72, 96,120h
Cmax of HGP1501 | 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72, 96,120h
baseline corrected AUCinf of HGP1501 | 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72, 96,120h
baseline corrected Tmax of HGP1501 | 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72, 96,120h
baseline corrected T1/2 of HGP1501 | 0,1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 48, 72, 96,120h

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Asan Hospital, Seoul, South Korea